CLINICAL TRIAL: NCT06311617
Title: Understanding Retinal Vascular Changes During Pregnancy and the Impact on Maternal and Fetal Health
Brief Title: Retinal Vascular Changes During Pregnancy
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Avni Finn, Principal Investigator, Medical Director of Imaging, Vanderbilt University Medical Center
Other Study IDs: 231592
Record Dates: First submitted 2024-03-02; First posted 2024-03-15 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy
Keywords: Optical coherence tomography; Pregnancy; Imaging; Retina; Vascular; Fundus Photography
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy Pregnant Patients: Health pregnancies
  Interventions: Diagnostic Test: Optical coherence tomography
- Pregnant Patients with Pre-Existing Diabetes: Patients with pre-existing diabetes who are pregnant
  Interventions: Diagnostic Test: Optical coherence tomography
- Pregnant Patients with Vascular Disease or Risk Factors for Vascular Disease: 1. Multiple gestations
  2. Preeclampsia or eclampsia
  3. Gestational diabetes
  4. Hypercoagulable state such as disseminated intravascular coagulation (DIC), thrombotic thrombocytopenic purpura (TTP), and hemolysis, elevated liver enzymes, and low platelets (HELLP) syndrome.
  Interventions: Diagnostic Test: Optical coherence tomography

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography — Non-mydriatic fundus photography and optical coherence tomography will be performed at 3 timepoints

SUMMARY:
The goal of this study is to better understand how the back part of the eye-called the retina and the choroid-changes during pregnancy. Specialized photos of the eye will be taken at three different timepoints: early in pregnancy (first or second trimester), late in pregnancy (third trimester), and after delivery. This imaging is non-invasive and does not require contact with the surface of the eye. The photos taken will allow assessment of specific parameters, like blood flow and the health of specialized cells that support vision. Understanding how the eyes change during pregnancy may help guide how retina specialists understanding of retinal disease during pregnancy and better inform pregnancy outcomes.

DETAILED DESCRIPTION:
Pregnancy is a unique human condition marked by changes throughout the body, including changes in hormone levels, blood volume, blood pressure, and blood clot formation. These changes impact the eye as well, particularly the back part of the eye, called the retina and the choroid. Pre-existing conditions like diabetes and high blood pressure are known to affect the retina, but this impact may be increased by during pregnancy. In addition, new eye conditions may develop. The purpose of this study is to better understand how the retina and choroid changes during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 18 years and older
2. Patient able to provide informed consent
3. Pregnant at time of enrollment and in the 1st or 2nd trimester of pregnancy

Exclusion Criteria:

1. Other ocular disease that prevents imaging (significant cataract or other media opacity)
2. Unable to comply with imaging or follow-up through duration of study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant patients
Study Population: Pregnant patients (healthy and those with pre-existing diabetes/hypertension, and those with pregnancy-associated hypertension and diabetes or multiple gestations)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Imaging Biomarkers: Choroid | during 9 months of pregnancy and in the 3 months after pregnancy
  Choroidal thickness
Imaging Biomarkers: Vessel density | during 9 months of pregnancy and in the 3 months after pregnancy
  Vessel density
Imaging Biomarkers: Foveal avascular zone (FAZ) | during 9 months of pregnancy and in the 3 months after pregnancy
  FAZ area

SECONDARY OUTCOMES:
Fetal Health: delivery | at time of birth
  Modality of delivery
Fetal Health | at time of birth
  weight of baby at birth

CONTACTS AND LOCATIONS:
Overall Officials: Avni P Finn, MD, MBA, Principal Investigator — Vanderbilt Eye Institute
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No